CLINICAL TRIAL: NCT01245296
Title: Early Versus Delayed Cord Clamping at Term: Outcomes in Swedish Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Umeå University (Other); Halmstad County Hospital (Other); County Council of Halland, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NATIBAR08
Record Dates: First submitted 2010-10-13; First posted 2010-11-22 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Iron Deficiency; Neonatal Hyperbilirubinemia
Keywords: Umbilical cord; cord clamping; iron; Ferritin; newborn; jaundice; infant; development; infections
MeSH Terms: conditions — Iron Deficiencies; Hyperbilirubinemia, Neonatal; Jaundice; Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early cord clamping (ECC) (Other): Early cord clamping consisted of early (< 10 s) clamping of the umbilical cord and obtaining blood gas samples after clamping.
  Interventions: Procedure: Timing of clamping the umbilical cord
- Delayed cord clamping (DCC) (Other): Delayed cord clamping consisted of delayed (> 180 s) clamping of the umbilical cord and obtaining blood gas samples before clamping (within 30 seconds).
  Interventions: Procedure: Timing of clamping the umbilical cord

INTERVENTIONS:
Procedure: Timing of clamping the umbilical cord — The time passed after delivery until that the midwife stops circulation in the umbilical cord with a clamp.
  Other Names: Delayed cord clamping is also called Late cord claming

SUMMARY:
Delayed clamping of the umbilical cord might prevent or slow the onset of iron deficiency by increasing the infant's iron endowment at birth. Compared with early clamping, a delay of around 2-3 min provides an additional 25-40 mL of blood per kg of bodyweight.

The results of previous intervention studies on delayed clamping are mixed, and few followed up infants beyond the perinatal period. All longer follow up studies have been performed in low income countries. The main objectives, therefore, was to assess whether delayed cord clamping improves hematological and iron status at 4 respective 12 months of age in a large sample of full-term, Swedish infants.

The investigators also choose to investigate if the timing of clamping the umbilical cord could affect rate of infections during the first four months of life and to assess the infants development at 4 and 12 months of age.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking mother
* healthy mother (no hemolytic disease, no treatment with any of the following drugs: anticonvulsants, antidepressants, thyroid hormone, insulin, chemotherapy or cortisone),
* normal pregnancy (no preeclampsia, no diabetes, no prolonged rupture of membranes or signs of infection)
* single birth, term pregnancy (gestational age 37 +0 until 41 +6 weeks + days)
* expected vaginal delivery with cephalic presentation
* mother should be able to master Swedish well enough to participate in the study
* mother should live close enough to the hospital to be ready to return for follow up after four months.

Exclusion Criteria:

* Serious congenital malformation, syndrome or other congenital disease that can affect the outcome measures

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 392 (Actual)
Dates: Start 2008-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Do time for clamping the umbilical cord affect children's hemoglobin and iron status at 4 months of age? | 4 months of age (plus or minus three weeks)
  Using mean cell volume (MCV), mean cell hemoglobin concentration (MCHC), reticulocyte hemoglobin, serum ferritin, transferrin saturation and soluble transferrin receptors to assess iron status

SECONDARY OUTCOMES:
Do the time for clamping the umbilical cord affect children's hemoglobin and iron status at 12 months of age? | 12 months of age (plus or minus one month)
  Using mean cell volume (MCV), mean cell hemoglobin concentration (MCHC), reticulocyte hemoglobin, serum ferritin, transferrin saturation and soluble transferrin receptors to assess iron status.
Are the rates of successful umbilical arterial samples equal between the groups? | Immediately after birth (within 30 seconds)
  Arterial blood samples are obtained with different methods between groups: in the early clamped group samples are taken from the placental part of the clamped cord, in the delayed clamped group samples are taken before clamping in the still pulsating cord. At the same time umbilical venous samples are obtained. A arterial blood sample is assessed as successful when ph < 0.2 and partial pressure of carbon dioxide (pCO2) > 0.5 kPa compared to the venous sample.
Is there a difference in development as assessed by the Ages and Stages Questionnaire at 4 months of age? | 4 months of age (plus or minus three weeks)
  Ages and Stages Questionnaire is a parent report questionnaire available for developmental screening of children from one month to 5 ½ years. 30 questions are divided into 5 developmental domains (communication, gross motor, fine motor, problem solving and personal-social). Total score and scores within separate domains from the 4-month questionnaire will be assessed.
Do the time for umbilical cord clamping affect incidence of infections during the first four months of life? | 4 months of age (plus or minus three weeks)
  After birth of their child, until four months of age parents fill out a form where they daily note if their infant has intestinal or respiratory symptoms, as well as if the infant has middle ear infection, has visited a doctor, has had an antibiotic prescription or has been admitted into a hospital.
Is Reticulocyte hemoglobin a useful measure of iron stores at 2-3 days of age? | Mean 2 to 3 days of age (within 48-96 hours after birth)
  Reticulocyte hemoglobin (RetHE) is a novel measure suggested to describe iron status. Ret HE will be compared to other indicators of iron stores: mean cell volume (MCV), mean cell hemoglobin concentration (MCHC), serum ferritin, transferrin saturation and soluble transferrin receptors
Do the time for umbilical cord clamping affect neonatal outcomes: anemia, polycythemia and need for phototherapy? | Within 7 days after birth
  Anemia defined as hemoglobin < 145 g/L, polycythemia defined as hematocrit > 0.65.
Is there any difference in post partum haemorrhage when using early cord clamping compared to delayed cord clamping with oxytocin administered after clamping? | After giving birth until discharge from maternity ward
  Measuring time to placental abortion, post partal hemorrhage and mothers post partum need for blood transfusion
Is there a difference in development as assessed by the Ages and Stages Questionnaire at 12 months of age? | 12 months of age (plus or minus one month)
  Ages and Stages Questionnaire is a parent report questionnaire available for developmental screening of children from one month to 5 ½ years. 30 questions are divided into 5 developmental domains (communication, gross motor, fine motor, problem solving and personal-social). Total score and scores within separate domains from the 12-month questionnaire will be assessed.
Do the time for umbilical cord clamping affect Immunoglobulin G levels at 2-3 days of age? | Mean 2 to 3 days of age (within 48-96 hours after birth)
  Blood samples for metabolic screening are routinely taken as soon as possible after 2 days (48 hours) of age. At the same time samples for Immunoglobulin G is obtained.
Is Reticulocyte hemoglobin a useful measure of iron stores at 12 months of age? | 12 months of age (plus or minus one month)
  Reticulocyte hemoglobin (RetHE) is a novel measure suggested to describe iron status. Ret HE will be compared to other indicators of iron stores: mean cell volume (MCV), mean cell hemoglobin concentration (MCHC), serum ferritin, transferrin saturation and soluble transferrin receptors
Does the time for umbilical cord clamping affect the infants respiration within the first 6 hours of life? | Within 6 hours after birth
  Midwives observes the newborn infant at 1 hour and 6 hours of age and note presence of tachypnea (> 60 breaths/minute), grunting, nostril flaring and or retractions between or under the ribs.

CONTACTS AND LOCATIONS:
Overall Officials: Ola Andersson, M.D., Principal Investigator — Uppsala University; Magnus Domellöf, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Länsjukhuset i Halmstad, Halmstad, Halland County, Sweden

REFERENCES:
- [Background] Begley CM, Gyte GM, Murphy DJ, Devane D, McDonald SJ, McGuire W. Active versus expectant management for women in the third stage of labour. Cochrane Database Syst Rev. 2010 Jul 7;(7):CD007412. doi: 10.1002/14651858.CD007412.pub2. PMID 20614458
- [Background] Chaparro CM, Fornes R, Neufeld LM, Tena Alavez G, Eguia-Liz Cedillo R, Dewey KG. Early umbilical cord clamping contributes to elevated blood lead levels among infants with higher lead exposure. J Pediatr. 2007 Nov;151(5):506-12. doi: 10.1016/j.jpeds.2007.04.056. Epub 2007 Sep 17. PMID 17961694
- [Background] Ceriani Cernadas JM, Carroli G, Pellegrini L, Otano L, Ferreira M, Ricci C, Casas O, Giordano D, Lardizabal J. The effect of timing of cord clamping on neonatal venous hematocrit values and clinical outcome at term: a randomized, controlled trial. Pediatrics. 2006 Apr;117(4):e779-86. doi: 10.1542/peds.2005-1156. Epub 2006 Mar 27. PMID 16567393
- [Background] van Rheenen P, de Moor L, Eschbach S, de Grooth H, Brabin B. Delayed cord clamping and haemoglobin levels in infancy: a randomised controlled trial in term babies. Trop Med Int Health. 2007 May;12(5):603-16. doi: 10.1111/j.1365-3156.2007.01835.x. PMID 17445128
- [Background] van Rheenen PF, Gruschke S, Brabin BJ. Delayed umbilical cord clamping for reducing anaemia in low birthweight infants: implications for developing countries. Ann Trop Paediatr. 2006 Sep;26(3):157-67. doi: 10.1179/146532806X120246. PMID 16925952
- [Background] Hutton EK, Hassan ES. Late vs early clamping of the umbilical cord in full-term neonates: systematic review and meta-analysis of controlled trials. JAMA. 2007 Mar 21;297(11):1241-52. doi: 10.1001/jama.297.11.1241. PMID 17374818
- [Background] Grajeda R, Perez-Escamilla R, Dewey KG. Delayed clamping of the umbilical cord improves hematologic status of Guatemalan infants at 2 mo of age. Am J Clin Nutr. 1997 Feb;65(2):425-31. doi: 10.1093/ajcn/65.2.425. PMID 9022526
- [Background] McDonald SJ, Middleton P. Effect of timing of umbilical cord clamping of term infants on maternal and neonatal outcomes. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD004074. doi: 10.1002/14651858.CD004074.pub2. PMID 18425897
- [Background] Mercer JS. Current best evidence: a review of the literature on umbilical cord clamping. J Midwifery Womens Health. 2001 Nov-Dec;46(6):402-14. doi: 10.1016/s1526-9523(01)00196-9. PMID 11783688
- [Result] Andersson O, Hellstrom-Westas L, Andersson D, Domellof M. Effect of delayed versus early umbilical cord clamping on neonatal outcomes and iron status at 4 months: a randomised controlled trial. BMJ. 2011 Nov 15;343:d7157. doi: 10.1136/bmj.d7157. PMID 22089242
- [Result] Andersson O, Domellof M, Andersson D, Hellstrom-Westas L. Effect of delayed vs early umbilical cord clamping on iron status and neurodevelopment at age 12 months: a randomized clinical trial. JAMA Pediatr. 2014 Jun;168(6):547-54. doi: 10.1001/jamapediatrics.2013.4639. PMID 24756128
- [Result] Andersson O, Domellof M, Andersson D, Hellstrom-Westas L. Effects of delayed cord clamping on neurodevelopment and infection at four months of age: a randomised trial. Acta Paediatr. 2013 May;102(5):525-31. doi: 10.1111/apa.12168. Epub 2013 Feb 11. PMID 23336628
- [Result] Andersson O, Hellstrom-Westas L, Andersson D, Clausen J, Domellof M. Effects of delayed compared with early umbilical cord clamping on maternal postpartum hemorrhage and cord blood gas sampling: a randomized trial. Acta Obstet Gynecol Scand. 2013 May;92(5):567-74. doi: 10.1111/j.1600-0412.2012.01530.x. Epub 2012 Oct 17. PMID 22913332
- [Derived] Askelof U, Andersson O, Domellof M, Fasth A, Hallberg B, Hellstrom-Westas L, Pettersson K, Westgren M, Wiklund IE, Gotherstrom C. Wait a minute? An observational cohort study comparing iron stores in healthy Swedish infants at 4 months of age after 10-, 60- and 180-second umbilical cord clamping. BMJ Open. 2017 Dec 29;7(12):e017215. doi: 10.1136/bmjopen-2017-017215. PMID 29289934